CLINICAL TRIAL: NCT05743478
Title: Forging Hopeful Futures: A Racial and Gender-Justice Program to Reduce Youth Violence
Brief Title: Forging Hopeful Futures to Reduce Youth Violence
Acronym: FHF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Population Council (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alison Culyba, Assistant Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY22080150; R01CE003502 (NIH)
Record Dates: First submitted 2023-02-13; First posted 2023-02-24 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Violence in Adolescence; Racism; Adolescent Behavior; Coping Skills; Communication, Social; Communication, Personal; Violence, Sexual; Violence, Non-accidental; Violence, Physical; Violence, Gender-Based
MeSH Terms: conditions — Racism; Adolescent Behavior; Communication; Coitus

STUDY DESIGN:
Intervention Model Description: This community-partnered cluster-randomized study will examine the effectiveness of a racial, gender, and economic justice focused youth violence prevention program called Forging Hopeful Futures among youth ages 13-19.The study will be located in 16 neighborhoods with concentrated disadvantage ('clusters') across Pittsburgh, Pennsylvania and urban Washington D.C. and Maryland metro areas randomized either to receive the "Forging Hopeful Futures" program (i.e., intervention neighborhood, n=8) or wellness check-ins (i.e. control neighborhood, n=8).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forging Hopeful Futures (Experimental): Forging Hopeful Futures uses a group discussion format with activities that explore race, gender, class, identity, relationships, and multiple forms of violence. Forging Hopeful Futures is a 12 session curriculum for youth ages 13-19 that uses strengths-based and healing-centered approaches to critically examine structural forces that perpetuate racial and gender injustice, develop leadership skills in promoting gender equitable relationship norms, non-violent practices, and upstander skills, and enhance economic justice through job skills and employment opportunities. Through 12 sessions (3 hours/session) over a 6 to 12 week period, Forging Hopeful Futures combines racial, gender, and economic justice content with leadership development and workforce development opportunities.
  Interventions: Behavioral: Forging Hopeful Futures
- Wellness Check-ins (Active Comparator): Youth in neighborhoods randomized to the control group will receive individual wellness checks. This will occur through a strengths-based telephone conversation focused on wellness resources. Youth will be provided with tailored resources based on needs identified during the call. Youth will be offered the option for additional phone check-ins to coordinate access to community resources and connection to individualized behavioral health supports if desired.
  Interventions: Behavioral: Wellness Check-ins

INTERVENTIONS:
Behavioral: Forging Hopeful Futures — Forging Hopeful Futures is a 12 session curriculum for youth ages 13-19 that uses strengths-based and healing-centered approaches to critically examine structural forces that perpetuate racial and gender injustice, develop leadership skills in promoting gender equitable relationship norms, non-violent practices, and upstander skills, and enhance economic justice through job skills and employment opportunities. Through 12 sessions (3 hours/session) over a 6 to 12 week period, Forging Hopeful Futures combines racial, gender, and economic justice content with leadership development and workforce development opportunities.
  Arms: Forging Hopeful Futures
Behavioral: Wellness Check-ins — Individual wellness checks will occur through a strengths-based telephone conversation focused on wellness resources. Youth will be provided with tailored resources based on needs identified during the call. Youth will be offered the option for additional phone check-ins to coordinate access to community resources and connection to individualized behavioral health supports if desired.
  Arms: Wellness Check-ins

SUMMARY:
This cluster-randomized community-partnered study will examine the effectiveness of a racial-, gender-, and economic-justice focused youth violence prevention program called Forging Hopeful Futures with youth ages 13-19.

DETAILED DESCRIPTION:
This community-partnered cluster randomized trial in 16 neighborhoods impacted by structural inequities and high levels of community violence in Pittsburgh, PA and urban Washington D.C. and Maryland metro areas will evaluate effectiveness of Forging Hopeful Futures with youth ages 13-19. Forging Hopeful Futures combines economic justice content from job readiness training, racial and gender justice content from gender-transformative programming, and leadership building as a novel multi-level violence prevention intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ages 13-19 (inclusive)
2. Participants must speak English
3. Participants must live in the participating neighborhoods, attend schools in the participating neighborhoods, or use participating facilities
4. Participants must be able to provide follow up contact information

Exclusion Criteria:

1. Not ages 13 -19 (inclusive)
2. Do not speak English
3. Do not live in the participating neighborhoods, attend schools in the participating neighborhoods, or use participating facilities
4. Unable to provide follow up contact information

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 720 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in recent violence perpetration at 3 months | At baseline and three months after program conclusion
  The primary outcome will be past 3-month youth violence perpetration. This will be measured by self-report on 3 items adapted from the Youth Risk Behavior Surveillance Survey, using a past-3 month reporting interval: 1) physical fighting ("How many times were you in a physical fight?"), 2) threatening someone with a weapon ("How many times have you threatened someone with a weapon such as a gun, knife, or club?"), and 3) injuring someone with a weapon ("How many times have you injured someone with a weapon such as a gun, knife, or club?"). Each item will be assessed with 8 frequency response categories from 0 times to 12 or more times. A summary score will capture the past 3-month incidence of all 3 behaviors (possible range: 0- 21;lower score indicates better outcome)

SECONDARY OUTCOMES:
Change in recent violence perpetration at 6 months | At baseline and six months after program conclusion
  This will be measured using the same 3 items outlined in the primary outcome, but assessed as a change from baseline to 6 months after program conclusion. This includes self-report on 3 items adapted from the Youth Risk Behavior Surveillance Survey, using a past-3 month reporting interval: 1) physical fighting ("How many times were you in a physical fight?"), 2) threatening someone with a weapon ("How many times have you threatened someone with a weapon such as a gun, knife, or club?"), and 3) injuring someone with a weapon ("How many times have you injured someone with a weapon such as a gun, knife, or club?"). Each item will be assessed with 8 frequency response categories from 0 times to 12 or more times. A summary score will capture the past 3-month incidence of all 3 behaviors (possible range: 0- 21;lower score indicates better outcome)
Change in relationship abuse at 3 months | At baseline and three months after program conclusion
  10 abusive behavior items, modified from Conflict Tactics Scale-2, assess for perpetration against dating partners or towards peers. Summary score of any recent use of violence in the past 3 months (physical, sexual and emotional relationship abuse) calculated as one point for each behavior then summed (possible range: 0-10; lower score indicates better outcome).
Change in sexual violence perpetration at 3 months | At baseline and three months after program conclusion
  4 sexual violence perpetration items assess recent sexual violence perpetration (any/none). Summary score of any recent sexual violence perpetration in the past 3 months, calculated as one point for each behavior then summed (possible range: 0-4; lower score indicates better outcome).
Change in cyber dating abuse and peer abuse | At baseline and three months after program conclusion
  8 items assess using technology to perpetrate abuse against a dating partner or peers. Summary score of any recent use of technology to perpetrate abuse against a dating partner or peers in the past 3 months, calculated as one point for each behavior then summed (possible range: 0-8; lower score indicates better outcome).
Change in bullying perpetration | At baseline and three months after program conclusion
  6 items to indicate frequency of bullying perpetration on 4-point frequency scale. Mean score of any recent bullying perpetration in the past 3 months, calculated as a mean score across the 6 items (possible range: 0-3; lower score indicates better outcome).
Change in cyberbullying perpetration | At baseline and three months after program conclusion
  4-item scale adapted from a cyberbullying perpetration scale, assessing perpetration frequency on a 4-point frequency scale. Mean score of recent cyberbullying perpetration in the past 3 months, calculated as a mean across the 4 items (possible range:0-3; lower score indicated better outcome).
Change in weapon carrying | At baseline and three months after program conclusion
  1 item adapted from the Youth Risk Behavior Surveillance Survey asking about frequency of carrying a weapon in the past 30 days (measured on a 5-point frequency scale from 0 days to 6 or more days; possible range: 0-4; lower score indicates better outcome).
Change in homophobic teasing | At baseline and three months after program conclusion
  5-item scale with participants reporting how often they have perpetrated listed behaviors in the past 3 months (each item measured on a 6-point frequency scale from 0 times to 7 or more times). Mean score of recent homophobic teasing, calculated as a mean across the 5 items (possible range: 0-5; lower score indicates better outcome).
Change in sexual harassment | At baseline and three months after program conclusion
  5 items assess frequency of perpetrating sexual harassing behaviors in the past 3 months, assessing perpetration frequency on a 5-point frequency scale. Mean score of recent sexual harassment perpetration in the past 3 months, calculated as a mean across the 5 items (possible range:0-4; lower score indicated better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Alison Culyba, MD PhD MPH, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Population Council, Washington D.C., District of Columbia
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
IDP data will be made available only to selected researchers who apply for access. The application must document a legitimate public health use or research question for the data, and the applicant must sign a pledge to keep all data private and to make no attempt to identify individual subjects. Access can be requested for all of the individual participant data collected during the trial, after deidentification. We will use data standards that ensure all released data have appropriate documentation that describes the method of collection, what the data represent, and potential limitations for use. Along with restricted use of the IDP, we will make available a comprehensive data dictionary that details all data elements included in the dataset, and sources of validated instruments. This use of the data is consistent with the planned language of the voluntary consent for participation agreed and in accordance with IRB policy.
Time Frame: We will adhere to data sharing timelines, including sharing data (restricted use) within 30 months after the end of data collection.
Access Criteria: We will make the data available only to selected researchers who apply for access. The application must document a legitimate public health use or research question for the data, and the applicant must sign a pledge to keep all data private and to make no attempt to identify individual subjects. This use of the data is consistent with the planned language of the voluntary consent for participation agreed and in accordance with IRB policy.